CLINICAL TRIAL: NCT04115280
Title: Prevalence of Primary Aldosteronism Among Hypertensive Patients Younger Than 65 Years Old With Atrial Arythmia
Brief Title: Prevalence of Primary Aldosteronism Among Hypertensive Patients With Atrial Arythmia
Acronym: HAPAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHPAU2019/01
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Primary Aldosteronism; Atrial Fibrillation
MeSH Terms: conditions — Hyperaldosteronism; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Primary Hyperaldosteronism diagnostic — blood sample to obtain the aldosterone to renin ratio

SUMMARY:
Atrial arrhythmia is the most frequent cardiac arrhythmia. It is a source of significant morbidity.

Hypertension is a major risk factor for atrial arrhythmias. Primary hyperaldosteronism (PA) is a common cause of secondary hypertension, associated with a high prevalence of arrhythmias with a specific, sometimes curative, treatment. The purpose of the study is to show that the prevalence of PA among hypertensive patients under 65 years old with atrial arrhythmia is high, justifying systematic screening.

DETAILED DESCRIPTION:
Atrial arrhythmia is the most frequent cardiac arrhythmia, affecting one million patients in France. It is a source of significant morbidity, a major deterioration in the quality of life and considerable health expenditure.

Hypertension is a major and modifiable risk factor for atrial arrhythmias. Primary hyperaldosteronism is a common cause of secondary hypertension, associated with a high prevalence of arrhythmias, but also stroke, coronary artery disease, heart and kidney failure. This form has a specific treatment, sometimes curative.

The objective of this study is to show that the prevalence of primary hyperaldosteronism among patients under 65 with atrial arrhythmias is high, justifying systematic screening in this population.

The investigators will consecutively include 65-year-old hypertensive patients hospitalized in the department with atrialarrhythmia. They will benefit from an aldosterone to renin ratio assay under standardized conditions at 3 months.

Patients whose aldosterone (pmol/l) to renin (mUI/l) ratio is greater than 64 will benefit from saline infusion test if necessary and adrenal scan. Patients with a definite diagnosis who would prefer surgical treatment will benefit from adrenal venous catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients aged of 18 to 65 years with atrial arrhythmia.

Exclusion Criteria:

* BMI above 30
* Any situation where the discontinuation of treatments (including betablockers and diuretics) presents a risk according to the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of the prevalence of primary hyperaldosteronism | Data collected after the saline infusion test (6-month visit)
  Prevalence of primary hyperaldosteronism among the enrolled population.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - CH de Pau, Pau

IPD SHARING:
Plan to Share IPD: No